CLINICAL TRIAL: NCT05777551
Title: Atrial Fibrillation Ablation by Means of Very High Power Short Duration (AIR HPSD Registry)
Brief Title: AF Ablation With High Power Short Duration RF
Acronym: AIR HPSD
Status: Recruiting | Type: Observational
Sponsor: Clinica Mediterranea (Other)
Responsible Party: Sponsor
Other Study IDs: AIR HPSD
Record Dates: First submitted 2023-02-15; First posted 2023-03-21 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Atrial Fibrillation; Catheter Ablation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a prospective, multi-center, research study designed to evaluate the safety and efficacy of pulmonary vein (PV) isolation with high power short duration radiofrequency energy in patients with paroxysmal/persistent atrial fibrillation (AF).

Subjects with paroxysmal/persistent AF will undergo catheter ablation using commercially approved devices (mapping system and catheters).

Patients will be followed up for 12 months to measure the recurrence of AF and its predictors. The primary endpoint will be to investigate the association between clinical and procedural characteristics and the efficacy and the safety of PVI performed with HPSD.

At least 850 consecutive will be enrolled to have an adequate statistical power for the analysis of the primary endpoint. We assume that the freedom form AF recurrence at 12 months will be 80%. Expected R^2 (Cox-Snell) 0.1. Candidate variables to be included in the model:10. Shrinkage level: 0.9. Based on these assumption the minimum number of patients is 850 with 170 events and EPP 17.

DETAILED DESCRIPTION:
Patients will be screened in ambulatory and scheduled for AF ablation according to current guidelines. Ablation will be usually performed under effective oral anticoagulation. Anticoagulation could be withdrawn before admission, so as antiarrhythmic drugs will be removed before scheduled procedure. Patients in AF or with a CHA2DS2-VASc score ≥ 1 will undergo transesophageal echocardiography within 48 hours prior to the ablation. For all other patients transesophageal echocardiography is optional. Cardiac MRI or Cardiac CT scan could be executed as a reference for volume estimations obtained with the mapping system.

Ablation will be carried out under mild or deep sedation, or general anesthesia according to center preference. At least 2 femoral vein access will be obtained and in some patients 1 subclavian vein. One diagnostic catheter will be positioned in the coronary sinus. One or two transseptal accesses to the left atrium will be achieved using a standard approach. Then, the mapping catheter (LASSO, Penta-ray, Octa-ray catheter) and the ablation catheter (QDot Micro catheter) will be placed in the left atrium. Heparin will be administered before the transseptal punctures to maintain an activated clotting time ≥ 300 seconds for the duration of the procedure. Left atrium mapping will be performed in sinus rhythm. Patients with atrial fibrillation at the beginning of the index procedure will undergo electrical cardioversion. After left atrium reconstruction the effective PV-left atrium electrical connection will be checked with the mapping catheter. In all patients a wide antrum circumferential ablation aimed at PV isolation will be performed using the QDot Micro catheter in QMode+ mode (90 w for 4 sec) for the whole ablation or in an hybrid mode (QMode + for posterior wall and QMode guided by AI in the anterior wall), according to the operator preference. The maximum interlesion distance will be <6 mm (16,17). According to operator preference it will be performed an ablation line encircling each PV or two ablation lines encircling the right and the left PVs. At the end of the ablation effective PV isolation (entry and exit block), will be checked with mapping catheter. After PV isolation will be achieved, the reconnection of the same vein will be evaluated after a 20 minute period from the initial isolation or after adenosine infusion or isoproterenol. If the vein reconnects to the atrium, the ablation will be directed to the gaps identified by the mapping catheter.

All patients will undergo a post-procedural ECG and, optional, an echocardiogram to exclude pericardial effusion or other acute complications.

After ablation, patients will undertake regular follow-up assessments (scheduled at 3 months) including a detailed history, physical examination, 12-lead standard electrocardiography, and 24-h Holter monitoring. Patients who will not report any symptoms related to the previous arrhythmia during a supplementary detailed follow up (6-12 months subsequent to catheter ablation) will be considered free of arrhythmia recurrence

ELIGIBILITY:
Inclusion Criteria:

* Patients with paroxysmal/persistent AF who signed the informed consent
* Patients on active oral anticoagulation

Exclusion Criteria:

* Previous ablation for AF
* Patients with LVEF<35%
* Women potentially pregnant
* Contraindications to X-ray exposure
* Congenital heart disease or cardiac surgery within 1 month

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with paroxysmal/persistent AF with indication to catheter ablation according to current guidelines
Sampling Method: Probability Sample
Enrollment: 850 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Association between clinical and procedural characteristics and the percentage of arrhythmia recurrence rate after PV isolation performed with HPSD. | 12 months after ablation
  to assess the efficacy of the procedure in terms of atrial arrhythmia recurrence-free rate (binary outcome), with a number of candidate predictors equal to 10

SECONDARY OUTCOMES:
Percentage of acute pulmonary vein reconnection reconnection | 20 minutes after ablation
  After PV isolation will be achieved, the reconnection of the same vein will be evaluated after a 20 minute period from the initial isolation or after adenosine infusion or isoproterenol.
Procedural time | during the procedure
  The Investigators will calculate the overall procedural time (min)
Percentage of patients with atrial arrhythmias recurrence during the blanking period | 3 months after ablation
  Number of patients with an atrial arrhythmia (atrial fibrillation, atrial tachycardia, atrial flutter) episode lasting at least 30 sec during the 3 month blanking period after the index ablation
Impact of anaesthesia type | during the procedure
  The Investigators will evaluate the type of anesthesia: (mild sedation, deep sedation, general anesthesia), the anesthetic drugs used and their dose in mg
Evaluation of pain perception during ablation | during the procedure
  The Investigators will assess the pain during the ablation with a 0-10 pain scale (0 no pain, 1-3 mild, 4-6 moderate, 7-9 severe, 10 very severe).
Fluoroscopy time | during the procedure
  The Investigators will calculate the overall fluoroscopy time (sec)
Radiofrequency time | during the procedure
  The Investigators will calculate the overall radiofrequency time (sec)

OTHER OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 30 days and 12 months after ablation
  Number of participants with treatment-related adverse events, acute and at 30-day and 12-month as assessed by CTCAE v4.0

CONTACTS AND LOCATIONS:
Locations (9):
- Centre Cardiologique Du Nord, Paris, France
- Italy (7):
  - Clinica Montevergine, Mercogliano, AV
  - Maria cecilia Hospital, Cotignola, RA
  - Ospedale di Conegliano, Conegliano, TV
  - Università Politecnica delle Marche, Ancona
  - Ospedale Civile di Asti, Asti
  - Clinica Mediterranea, Napoli
  - Città della Salute e della Scienza di Torino, Dipartimento di Scienze Mediche della Università di Torino., Torino
- Royal Papworth Hospital, Cambridge, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
all collected IPD
Supporting Information: Study Protocol, SAP, ICF
Time Frame: starting 6 months after publication on primary end point
Access Criteria: The data will be shared on reasonable request to the corresponding author

REFERENCES:
- [Result] Stabile G, Lepillier A, De Ruvo E, Scaglione M, Anselmino M, Sebag F, Pecora D, Gallagher M, Rillo M, Viola G, Rossi L, De Santis V, Landolina M, Castro A, Grimaldi M, Badenco N, Del Greco M, De Simone A, Pisano E, Abbey S, Lamberti F, Pani A, Zucchelli G, Sgarito G, Dugo D, Bertaglia E, Strisciuglio T, Solimene F. Reproducibility of pulmonary vein isolation guided by the ablation index: 1-year outcome of the AIR registry. J Cardiovasc Electrophysiol. 2020 Jul;31(7):1694-1701. doi: 10.1111/jce.14531. Epub 2020 May 11. PMID 32369225
- [Result] Duytschaever M, Vijgen J, De Potter T, Scherr D, Van Herendael H, Knecht S, Kobza R, Berte B, Sandgaard N, Albenque JP, Szeplaki G, Stevenhagen YJ, Taghji P, Wright M, Macours N, Gupta D. Standardized pulmonary vein isolation workflow to enclose veins with contiguous lesions: the multicentre VISTAX trial. Europace. 2020 Nov 1;22(11):1645-1652. doi: 10.1093/europace/euaa157. PMID 32879974
- [Result] Ouyang F, Antz M, Ernst S, Hachiya H, Mavrakis H, Deger FT, Schaumann A, Chun J, Falk P, Hennig D, Liu X, Bansch D, Kuck KH. Recovered pulmonary vein conduction as a dominant factor for recurrent atrial tachyarrhythmias after complete circular isolation of the pulmonary veins: lessons from double Lasso technique. Circulation. 2005 Jan 18;111(2):127-35. doi: 10.1161/01.CIR.0000151289.73085.36. Epub 2004 Dec 27. PMID 15623542
- [Result] Lemola K, Hall B, Cheung P, Good E, Han J, Tamirisa K, Chugh A, Bogun F, Pelosi F Jr, Morady F, Oral H. Mechanisms of recurrent atrial fibrillation after pulmonary vein isolation by segmental ostial ablation. Heart Rhythm. 2004 Jul;1(2):197-202. doi: 10.1016/j.hrthm.2004.03.071. PMID 15851153
- [Result] Cappato R, Negroni S, Pecora D, Bentivegna S, Lupo PP, Carolei A, Esposito C, Furlanello F, De Ambroggi L. Prospective assessment of late conduction recurrence across radiofrequency lesions producing electrical disconnection at the pulmonary vein ostium in patients with atrial fibrillation. Circulation. 2003 Sep 30;108(13):1599-604. doi: 10.1161/01.CIR.0000091081.19465.F1. Epub 2003 Sep 8. PMID 12963643
- [Result] Wang XH, Liu X, Sun YM, Gu JN, Shi HF, Zhou L, Hu W. Early identification and treatment of PV re-connections: role of observation time and impact on clinical results of atrial fibrillation ablation. Europace. 2007 Jul;9(7):481-6. doi: 10.1093/europace/eum101. Epub 2007 May 23. PMID 17522081
- [Result] McLellan AJ, Kumar S, Smith C, Morton JB, Kalman JM, Kistler PM. The role of adenosine following pulmonary vein isolation in patients undergoing catheter ablation for atrial fibrillation: a systematic review. J Cardiovasc Electrophysiol. 2013 Jul;24(7):742-51. doi: 10.1111/jce.12121. Epub 2013 Mar 14. PMID 23489944
- [Result] Leshem E, Zilberman I, Tschabrunn CM, Barkagan M, Contreras-Valdes FM, Govari A, Anter E. High-Power and Short-Duration Ablation for Pulmonary Vein Isolation: Biophysical Characterization. JACC Clin Electrophysiol. 2018 Apr;4(4):467-479. doi: 10.1016/j.jacep.2017.11.018. Epub 2018 Feb 2. PMID 30067486
- [Result] Barkagan M, Contreras-Valdes FM, Leshem E, Buxton AE, Nakagawa H, Anter E. High-power and short-duration ablation for pulmonary vein isolation: Safety, efficacy, and long-term durability. J Cardiovasc Electrophysiol. 2018 Sep;29(9):1287-1296. doi: 10.1111/jce.13651. Epub 2018 Jun 20. PMID 29846987
- [Result] Reddy VY, Grimaldi M, De Potter T, Vijgen JM, Bulava A, Duytschaever MF, Martinek M, Natale A, Knecht S, Neuzil P, Purerfellner H. Pulmonary Vein Isolation With Very High Power, Short Duration, Temperature-Controlled Lesions: The QDOT-FAST Trial. JACC Clin Electrophysiol. 2019 Jul;5(7):778-786. doi: 10.1016/j.jacep.2019.04.009. Epub 2019 May 8. PMID 31320006
- [Result] Stabile G, Schillaci V, Strisciuglio T, Arestia A, Agresta A, Shopova G, De Simone A, Solimene F. In vivo biophysical characterization of very high power, short duration, temperature-controlled lesions. Pacing Clin Electrophysiol. 2021 Oct;44(10):1717-1723. doi: 10.1111/pace.14358. Epub 2021 Sep 15. PMID 34498748
- [Result] Halbfass P, Wielandts JY, Knecht S, Le Polain de Waroux JB, Tavernier R, De Wilde V, Sonne K, Nentwich K, Ene E, Berkovitz A, Mueller J, Lehmkuhl L, Reichart A, Lusebrink U, Duytschaever M, Deneke T. Safety of very high-power short-duration radiofrequency ablation for pulmonary vein isolation: a two-centre report with emphasis on silent oesophageal injury. Europace. 2022 Mar 2;24(3):400-405. doi: 10.1093/europace/euab261. PMID 34757432
- [Result] Richard Tilz R, Sano M, Vogler J, Fink T, Saraei R, Sciacca V, Kirstein B, Phan HL, Hatahet S, Delgado Lopez L, Traub A, Eitel C, Schluter M, Kuck KH, Heeger CH. Very high-power short-duration temperature-controlled ablation versus conventional power-controlled ablation for pulmonary vein isolation: The fast and furious - AF study. Int J Cardiol Heart Vasc. 2021 Jul 26;35:100847. doi: 10.1016/j.ijcha.2021.100847. eCollection 2021 Aug. PMID 34381869
- [Result] Sallo Z, Perge P, Balogi B, Orban G, Piros K, Herczeg S, Nagy KV, Osztheimer I, Abraham P, Merkely B, Geller L, Szegedi N. Impact of High-Power and Very High-Power Short-Duration Radiofrequency Ablation on Procedure Characteristics and First-Pass Isolation During Pulmonary Vein Isolation. Front Cardiovasc Med. 2022 Jul 7;9:935705. doi: 10.3389/fcvm.2022.935705. eCollection 2022. PMID 35872909
- [Result] Hindricks G, Potpara T, Dagres N, Arbelo E, Bax JJ, Blomstrom-Lundqvist C, Boriani G, Castella M, Dan GA, Dilaveris PE, Fauchier L, Filippatos G, Kalman JM, La Meir M, Lane DA, Lebeau JP, Lettino M, Lip GYH, Pinto FJ, Thomas GN, Valgimigli M, Van Gelder IC, Van Putte BP, Watkins CL; ESC Scientific Document Group. 2020 ESC Guidelines for the diagnosis and management of atrial fibrillation developed in collaboration with the European Association for Cardio-Thoracic Surgery (EACTS): The Task Force for the diagnosis and management of atrial fibrillation of the European Society of Cardiology (ESC) Developed with the special contribution of the European Heart Rhythm Association (EHRA) of the ESC. Eur Heart J. 2021 Feb 1;42(5):373-498. doi: 10.1093/eurheartj/ehaa612. No abstract available. PMID 32860505
- [Result] Park CI, Lehrmann H, Keyl C, Weber R, Schiebeling J, Allgeier J, Schurr P, Shah A, Neumann FJ, Arentz T, Jadidi AS. Mechanisms of pulmonary vein reconnection after radiofrequency ablation of atrial fibrillation: the deterministic role of contact force and interlesion distance. J Cardiovasc Electrophysiol. 2014 Jul;25(7):701-8. doi: 10.1111/jce.12396. Epub 2014 Apr 2. PMID 24575734
- [Result] Phlips T, Taghji P, El Haddad M, Wolf M, Knecht S, Vandekerckhove Y, Tavernier R, Duytschaever M. Improving procedural and one-year outcome after contact force-guided pulmonary vein isolation: the role of interlesion distance, ablation index, and contact force variability in the 'CLOSE'-protocol. Europace. 2018 Nov 1;20(FI_3):f419-f427. doi: 10.1093/europace/eux376. PMID 29315411